CLINICAL TRIAL: NCT02631317
Title: Hospital Processes Reengineering of Intravenous Thrombolysis in Acute Ischemic Stroke in China
Acronym: PROMISE
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, Anding Xu, Professor, First Affiliated Hospital of Jinan University
Other Study IDs: 2011BAI08B02-02
Record Dates: First submitted 2014-10-26; First posted 2015-12-16 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Ischemic Stroke; Adverse Effect of Thrombolytic Drugs, Sequela
Keywords: acute ischemic stroke; intravenous rt-PA thrombolysis; process reengineering; door-to-needle time
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- rt-PA: patients treated with rt-PA, followed strategies were used: advance hospital notification by EMS, stroke team notification, key performance indicators feedback form, standard informed consent procedures, performance of thrombolysis at CT-room.
  Interventions: Behavioral: Advance hospital notification by EMS; Behavioral: stroke team notification; Behavioral: key performance indicators feedback form; Behavioral: standard informed consent procedures; Behavioral: performance of thrombolysis at CT-room

INTERVENTIONS:
Behavioral: Advance hospital notification by EMS — Advance hospital notification by EMS
Behavioral: stroke team notification — stroke team notification
Behavioral: key performance indicators feedback form — a "key performance indicators real-time feedback form" as continuing quality improvement
Behavioral: standard informed consent procedures — standard informed consent procedures with public poster of thrombolysis
Behavioral: performance of thrombolysis at CT-room — performance of thrombolysis at CT-room or emergency room

SUMMARY:
PROMISE is a prospective, nationwide, multicenter, longitudinal cohort study, focusing on hospital intravenous thrombolysis process reengineering for acute ischemic stroke (AIS). With a proposed "Reengineered Process Framework" for intravenous thrombolysis process by the PROMISE study steering committee, about 30 medical centers enters would be recruited nationwide, and each center would include consecutive AIS patients with an onset-to-door time (ODT) of less than 3.5 h. The investigators hypothesize that the proposed "Reengineered Process Framework" is suitable and feasible for hospitals in mainland of China; the rate of intravenous rt-PA thrombolysis in ischemic stroke patients with an ODT of less than 3.5 h would be more than 20% or be increased by 40% as compared with baseline; the proportion of patients with a door-to-needle (DNT) time of less than 60 min would be more than 20%, or be with an increase by ≥ 40% as compared with baseline.

DETAILED DESCRIPTION:
1. After reviewing domestic and international clinical research literature, the PROMISE study steering committee constructed the "Reengineered Process Framework" for intravenous thrombolysis process with business process reengineering theory. The suggested "Reengineered Process Framework" is regarded as feasible and suitable for hospitals in mainland of China.
2. The study period is 12 months, of which the first 3 months is the baseline period. After 3 months, all centers should develop new thrombolytic processes according to the "Reengineered Process Framework". The new processes are gradually implemented since the 4th month with continues care quality improvements.
3. The "Reengineered Process Framework" adopts a form of comprehensive package, proposes unified key points of process reengineering, provides a series of supporting, standardized tools for process management, and establishes a real-time key performance indicator (KPI) monitoring feedback system, etc.
4. Supporting, standardized tools includes: rapid identification tools of suspected stroke for medical personnel in the emergency system; stroke team building programs; real-time feedback form of KPI; standardized thrombolysis informed consent form and informed conversation public service advertising posters; suggested indications and contraindications for intravenous thrombolysis; standard operation procedure of intravenous rt-PA thrombolysis, etc.

With these methods, it is expected to raise the thrombolytic rate for patients arrived at medical center within 3.5 hours after the onset, and to shorten the door to needle time in China.

ELIGIBILITY:
Inclusion Criteria:

* All AIS patients with an onset-to-door time of less than 3.5 h of onset; informed consent

Exclusion Criteria:

1. Complete remission of symptoms and signs, in consideration for patients with transient ischemic attack;
2. Silent cerebral infarction without symptoms or signs;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AIS patients with an onset-to-door time of less than 3.5 h
Sampling Method: Non-Probability Sample
Enrollment: 2178 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The thrombolysis rate of patients treated with rt-PA | within 4.5 hours
  The rate of intravenous rt-PA thrombolysis in ischemic stroke patients with an ODT of less than 3.5 h: ≥ 20%, with an increase over the baseline ≥ 40%
The rate of DNT less than 60 min within the patients treated with rt-PA | within 4.5 hours
  The rate of patients with a door-to-needle (DNT) time of less than 60 min for intravenous rt-PA thrombolysis: ≥20%, with an increase over the baseline ≥ 40%

SECONDARY OUTCOMES:
intravenous rt-PA thrombolysis with an ODT of less than 2 h | 3 hours
  intravenous rt-PA thrombolysis in ischemic stroke patients with an onset-to-door time(ODT) of less than 2 h
death or dependence at 3-month | 90 days
  "death or dependence at 3-month" was defined as modified Rankin Scale(mRS) score 3-6 points.
favorable outcome at 3-month | 90 days
  "favorable outcome at 3-month" was defined as mRS 0-1 points.

CONTACTS AND LOCATIONS:
Overall Officials: ANDING XU, Prof, Study Chair — Stroke Center, The First Affiliated Hospital,Jinan University Guanzghou